CLINICAL TRIAL: NCT03159104
Title: Multicenter Double-blind Placebo-Controlled Randomized Clinical Trial of Efficacy and Safety of Tenoten for Children in the Treatment of Specific Developmental Disorders of Scholastic Skills in Children
Brief Title: Efficacy and Safety of Tenoten for Children in the Treatment of Specific Developmental Disorders of Scholastic Skills in Children
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Materia Medica Holding (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MMH-TD-005
Record Dates: First submitted 2017-05-17; First posted 2017-05-18 (Actual); Results first posted 2023-08-21 (Actual); Last update posted 2023-08-21 (Actual); Status verified 2021-10

CONDITIONS: Specific Developmental Disorders of Scholastic Skills
MeSH Terms: interventions — tenoten

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tenoten for children (Experimental): Dose per administration: 1 tablet. 1 tablet three times daily (3 tablets per day). The tablets should be held in the mouth until complete dissolution, without meal.
  Interventions: Drug: Tenoten for children
- Placebo (Placebo Comparator): Dose per administration: 1 tablet. 1 tablet three times daily (3 tablets per day). The tablets should be held in the mouth until complete dissolution, without meal.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tenoten for children — Tablet for oral use.
  Arms: Tenoten for children
Drug: Placebo — Tablet for oral use.
  Arms: Placebo

SUMMARY:
Purpose of the study:

• To evaluate efficacy and safety of Tenoten for children in the treatment of specific developmental disorders of scholastic skills in children.

DETAILED DESCRIPTION:
A multicenter, double-blind, randomized, placebo-controlled clinical trial to evaluate the efficacy and safety of the study treatment.

The study will enroll the school children (boys and girls) of grades 1, 2 and 3 of a regular school aged 7-9 years old (grade 1 school children will be enrolled at the beginning of the second half of the year) complaining of difficult learning classified according to ICD-10 as specific developmental disorders of scholastic skills (F81) including:

* specific reading disorder (F81.0);
* specific spelling disorder (F81.1);
* specific disorder of arithmetical skills (F81.2);
* mixed disorder of scholastic skills (F81.3);
* disorder simultaneously meeting criteria of F81.2+F81.0 or F81.2+F81.1, or F81.2+F81.0+F81.1.

The developmental disorders of scholastic skills will be verified by a doctor (either a neurologist or psychiatrist) according to reading, spelling, and counting tests. The children may have any concomitant diseases not considered as exclusion criteria and not requiring therapy during the following 12 weeks using the products specified in section "Forbidden concomitant therapy". Specific additional educational programs should not be performed within 12 weeks after enrollment either.

On signing information sheet (informed consent form) by the parent/adopter the patients will be examined by a neurologist or psychiatrist and tested for reading skills (method by L.A. Fotekova, Т.V. Akhutina, 2002;), spelling skills (method by L.A. Fotekova, Т.V. Akhutina, 2002) and counting skills (subtest No. 3 "Arithmetic" WISC test), and concomitant therapy will be recorded.

If inclusion criteria are met and non-inclusion criteria are absent at Visit 1, the patient will be enrolled in the trial and randomized into one of the two groups: 1 tablet of Tenoten for children three times daily for 3 months (group 1) or the same dosing regimen of Placebo (group 2).

At Visit 1 the parents/adopters will receive the study product for 12-week treatment period and a diary to report any potential adverse events and cases of concomitant therapy.

Six weeks later (Week 6±3 days) a "Phone visit" (Visit 2) will be made in order to interview parents about the patient's condition, the presence/absence of concomitant diseases, adverse events.

At Visit 3 (Week 12±3 days) repeated testing of reading, spelling and counting skills will be made, complaints, data on concomitant diseases, concomitant therapy, and adverse events will be collected. The investigator will evaluate the subject's compliance and fill in the Clinical Global Impression Scale to calculate Efficacy Index (CGI-EI).

The patients will be allowed to take symptomatic therapy and medications for their co-morbidities during the study, except for the medicines listed in "Forbidden concomitant therapy".

ELIGIBILITY:
Inclusion Criteria:

1. Children of either gender aged 7 to 9 years old.
2. School children of grades 1-3 (grade 1 children will be enrolled at the beginning of the second half of the year) in regular schools with state accreditation with principal educational program of elementary general education in compliance with Federal State Educational Standard of the Russian Federation.
3. Beginning of the second half of the year (only for 1st grades).
4. Specific developmental disorder of scholastic skills such as:

   * specific reading disorder (F81.0);
   * specific spelling disorder (F81.1);
   * specific disorder of arithmetical skills (F81.2);
   * mixed disorder of scholastic skills (F81.3; i.e. meeting the criteria for one of the following combinations: F81.2+F81.0, F81.2+F81.1, or F81.2+F81.0+F81.1).
5. Reading score of 15 to 35 on the Reading Skills test (L.A. Fotekova, T.V. Akhutina, 2002).
6. Spelling score of 15 to 30 on the Spelling Skills test (L.A. Fotekova, T.V. Akhutina, 2002).
7. Counting score of 5 to 15 on subtest No. 3 "Arithmetic" (of Wechsler Intelligence Scale for Children).
8. Availability of a patient information sheet (Informed Consent form) signed by the parent/adopter to confirm the child's participation in the clinical trial.

Exclusion Criteria:

1. History of the diseases:

   * Diseases of the nervous system, including

     * inflammatory diseases of the central nervous system;
     * systemic atrophies;
     * extrapyramidal and movement disorders;
     * degenerative diseases of the nervous system;
     * demyelinating diseases of the central nervous system;
     * episodic and paroxysmal disorders;
     * polyneuropathies;
     * diseases of myoneural junction and muscle;
     * cerebral palsy.
   * Congenital malformations of the nervous system (excl. Spina bifida without hydrocephalus)
   * Diseases and congenital malformations of the eye causing impairment of vision.
   * Diseases and congenital malformations of the ear causing impairment of hearing.
   * Organic mental disorders.
   * Mental retardation ranging from mild to profound.
   * Stuttering (stammering).
   * Obsessive-compulsive disorder.
   * Pervasive developmental disorders including:

     * childhood autism;
     * atypical autism;
     * Rett syndrome;
     * overactive disorder associated with mental retardation and stereotyped movements;
     * Asperger syndrome.
   * Phakomatoses (tuberous sclerosis, neurofibromatosis).
   * Postconcussional syndrome.
   * Hereditary metabolic diseases, including glycogen storage disease (glycogenosis), disorders of galactose metabolism (galactosemia), other disorders of carbohydrate metabolism, disorders of glycosaminoglycan metabolism (mucopolysaccharidoses), disorders of aromatic amino-acid metabolism (phenylketonuria, tyrosinemia, etc.), disorders of branched-chain amino-acid metabolism and fatty-acid metabolism (maple-syrup-urine disease), mitochondrial myopathy.
   * Chromosomal abnormalities.
2. Administration of the products specified in section "Forbidden concomitant therapy" within the previous 4 weeks.
3. Necessity in pharmacotherapy for underlying and/or concomitant disease during the following 12 weeks.
4. Acute infectious disease or exacerbation/decompensation of a disease affecting the patient's ability to participate in the trial.
5. Malignant neoplasm/suspected malignant neoplasm.
6. Allergy/intolerance to any of the components of medications used in the treatment.
7. Malabsorption syndrome including congenital or acquired lactase deficiency (or another disaccharidase deficiency), and galactosemia.
8. Mental disorders of patient's parent(s)/adopter(s).
9. Use of drugs or alcohol by the patient's parents/adopters at > 2 alcohol units a day (1 unit of alcohol is equivalent to 0.33 L of lager/150 mL of unfortified wine, or 40 mL of Ethyl Alcohol).
10. Participation in other clinical trials in the previous 3 months.
11. Patients whose parent(s)/adopter(s), from the investigator's point of view, will fail to comply with the observation requirements of the trial or with the dose regimen of the investigational drug.
12. Patients whose parent(s)/adopter(s) are related to any of the on-site research personnel directly involved in the conduct of the trial or are an immediate relative of the study investigator. "Immediate relative" means husband, wife, parent, son, daughter, brother, or sister (regardless of whether they are natural or adopted).
13. Patients whose parent(s)/adopter(s) work for OOO "NPF "MATERIA MEDICA HOLDING" (i.e., is the company's employee, temporary contract worker, or, designated officials responsible for carrying out the research or any immediate relatives of the aforementioned).

Ages: 7 Years to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 240 (Actual)
Dates: Start 2015-08-25 (Actual); Primary Completion 2019-02-18 (Actual); Study Completion 2019-02-18 (Actual)

CONTACTS AND LOCATIONS:
Locations (10):
- Russia (10):
  - Federal State Budgetary Educational Institution of Higher Education "Kazan Medical University" of the Ministry of Healthcare of the Russian Federation, Kazan'
  - The State Budgetary Healthcare Institution "Specialized Clinical Psychiatric Hospital No. 1" of the Krasnodar Region Health Department, Krasnodar
  - Federal State Budgetary Educational Institution of Higher Education "Pirogov Russian National Research Medical University" of the Ministry of Healthcare of the Russian Federation, Moscow
  - Moscow Regional Research and Clinical Institute ("MONIKI"), Moscow
  - Limited Liability Company "NIZHMEDCLINIKA", Nizhny Novgorod
  - LLC City Neurological Center "Sibneyromed", Novosibirsk
  - Municipal budgetary health care institution "Children's City Polyclinic № 4 of Rostov-on-Don", Rostov-on-Don
  - St. Petersburg State Budgetary Institution of Health "Children's City Polyclinic № 35", Saint Petersburg
  - Pediatric Research and Clinical Center for Infectious Diseases, Saint Petersburg
  - State Budgetary Healthcare Institution of Sverdlovsk Region Children's Clinical Hospital of Rehabilitation The Scientific and Practical Center "Bonum", Yekaterinburg

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Tenoten for Children | Placebo
Started | 122 | 118
Completed | 121 | 116
Not Completed | 1 | 2
Not completed — Violation of inclusion criteria | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tenoten for Children | Placebo | Total
Number analyzed (Participants) | 121 | 116 | 237
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 121 | 116 | 237
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 8.5 (0.7) | 8.6 (0.6) | 8.6 (0.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 49 | 46 | 95
  Male | 72 | 70 | 142
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Russia | 121 | 116 | 237

OUTCOME MEASURES:

1. Primary Outcome: Mean Total Scholastic Skills Score (a Sum of Three Scales: Reading, Spelling, and Counting).
Description: The total scholastic skill score is calculated based on the points for reading, spelling, and counting skills.
  Reading skills are estimated according to scale consisting of three subscales:reading speed, reading method/understanding, and reading accuracy. The minimum value of reading skills scale is 0 points, and the maximum value is 45 points.
  Spelling skills are estimated according to scale in 0, 15, 30, and 45 points. The minimum value is 0 points, and the maximum value is 45 points.
  Counting skills are estimated according to subtest No. 3 "Arithmetic" of "Wechsler Intelligence Scale for Children" (WISC) in points. The minimum value is 0 points, and the maximum value is 20 points.
  Total scholastic skill score is a sum of three scales (reading, spelling, and counting). The minimum value is 0 points, and the maximum value is 110 points. A higher score means the best results.
Time Frame: On Day 1 and after 12 weeks of the therapy
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Tenoten for Children | Placebo
Number analyzed (Participants) | 121 | 116
score on a scale
  Baseline | 61.39 (12.04) | 60.46 (11.04)
  After 12 weeks | 79.94 (18.22) | 74.56 (18.75)
Statistical Analysis 1: Comparison: Tenoten for Children vs Placebo; The difference between final and initial total scholastic skill score was calculated for each participant. Wilcoxon test was used for comparison of these differences because data distribution differs from normal; Test type: Superiority; p = 0.0113, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = 5, 95% CI 2-sided [1 to 9] — Hodges-Lehmann estimator was used for the difference between median change of total scholastic skill score in each comparison group

2. Secondary Outcome: Mean Reading Skills Score
Description: Reading skills are estimated according to scale consisting of three subscales: reading speed, reading method/understanding, and reading accuracy.
  Students of 7 years old are invited to read the words, and students of 8-9 years old are invited to read a small text. Speed, method, and accuracy of the reading are estimated in students of 7 years old. Speed, accuracy, and understanding of the text are estimated in students of 8-9 years old.
  The minimum value is 0 points, and the maximum value is 45 points. A higher score meant the best results.
Time Frame: On Day 1 and after 12 weeks of the therapy
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Tenoten for Children | Placebo
Number analyzed (Participants) | 121 | 116
score on a scale
  Baseline | 27.69 (6.52) | 27.76 (6.16)
  After 12 weeks | 34.96 (6.66) | 33.66 (7.7)
Statistical Analysis 1: Comparison: Tenoten for Children vs Placebo; Test type: Superiority; p = 0.0608, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = 0, 95% CI 2-sided [0 to 5] — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Mean Score Spelling Skills Score
Description: Spelling skills are estimated according to scale in 0, 15, 30, and 45 points. Students of 7 years old are invited to write dictated letters, their names, and three words (mom, table, trunk), and students of 8-9 years old are invited to write a small dictation.
  Dysgraphic errors and their types as well as the number of non-dysgraphic errors are taken into consideration for estimation.
  The minimum value is 0 points, and the maximum value is 45 points. A higher score meant the best results.
Time Frame: On Day 1 and after 12 weeks of the therapy
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Tenoten for Children | Placebo
Number analyzed (Participants) | 121 | 116
score on a scale
  Baseline | 22.56 (7.53) | 21.59 (7.48)
  After 12 weeks | 32.73 (13.69) | 29.09 (14.58)
Statistical Analysis 1: Comparison: Tenoten for Children vs Placebo; Test type: Superiority; p = 0.0824, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = 0, 95% CI 2-sided [0 to 0] — [estimate comment as in outcome 1, analysis 1]

4. Secondary Outcome: Mean Counting Skills Score.
Description: Counting skills are estimated according to subtest No. 3 "Arithmetic" of "Wechsler Intelligence Scale for Children" (WISC) in points. "Arithmetic" subtest includes 16 tasks from elementary school arithmetic which are tackled verbally. Easiness of operating numbers, accuracy, and time spent on the tasks are estimated. Each task is rated in points (0 or 1), by the end of testing and rating for each task the sum of points (raw score) is calculated and converted into a scale score using standard tables.
  The minimum value is 0 points, and the maximum value is 20 points. A higher score meant the best results.
Time Frame: On Day 1 and after 12 weeks of the therapy
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Tenoten for Children | Placebo
Number analyzed (Participants) | 121 | 116
score on a scale
  Baseline | 11.14 (2.24) | 11.10 (2.27)
  After 12 weeks | 12.26 (2.80) | 11.80 (2.73)
Statistical Analysis 1: Comparison: Tenoten for Children vs Placebo; Test type: Superiority; p = 0.2391, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = 0, 95% CI 2-sided [0 to 1] — [estimate comment as in outcome 1, analysis 1]

5. Secondary Outcome: Percentage of Children With an Increase in Total Scholastic Skills Score (a Sum of Three Scales: Reading, Spelling, and Counting).
Description: Percentage of children with an increase in total scholastic skills score (a sum of three scales: reading, spelling, and counting).
  Total scholastic skill score is a sum of three scales (reading, spelling, and counting).
  The minimum value is 0 points, and the maximum value is 110 points. A higher score meant the best results. The increase in total scholastic skills score means an increasing by at least 5 points compared to baseline.
Time Frame: On Day 1 and after 12 weeks of the therapy
Measure: Count of Participants; unit: Participants
Arm/Group | Tenoten for Children | Placebo
Number analyzed (Participants) | 121 | 116
Participants | 103 | 80
Statistical Analysis 1: Comparison: Tenoten for Children vs Placebo; Test type: Superiority; p = 0.0033, Fisher Exact

6. Secondary Outcome: Efficacy Index According to Clinical Global Impression Scale.
Description: The Clinical Global Impression-Efficiency Index (CGI-E) scale consists of two subscales.
  Efficacy subscale measures efficacy of medicine based on the severity of symptoms at the end of therapy. The minimum value is 1 points, and the maximum value is 4 points. A higher score means the best results.
  Side effects subscale measures side effects of the medicine. The minimum value is 1 points, and the maximum value is 4 points. A higher score means the best results.
  The scale is filled in by the doctor at the final visit after 12 weeks of the treatment. In accordance with the results of treatment, the doctor expresses his opinion about the efficacy of the therapy and the degree of medicine safety, making marks in the appropriate columns of the table. The efficacy index is determined as intersection of columns of indicators of efficacy and side effects in the table. The minimum value is 0.25 points, and the maximum value is 4 points. A higher score means the best results.
Time Frame: In 12 weeks of the treatment.
Population: The number of patients who have data on the CGI-EI scale is indicated.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Tenoten for Children | Placebo
Number analyzed (Participants) | 118 | 112
score on a scale | 2.36 (0.87) | 1.98 (0.83)
Statistical Analysis 1: Comparison: Tenoten for Children vs Placebo; Test type: Superiority; p = 0.0012, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: During the treatment period - 12 weeks.
Arm/Group | Tenoten for Children | Placebo
All-Cause Mortality (participants affected / at risk) | 0/122 | 0/118
Serious Adverse Events (participants affected / at risk) | 0/122 | 2/118
Other Adverse Events (participants affected / at risk) | 42/122 | 29/118
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tenoten for Children (N=122) | Placebo (N=118)
Phlegmonous appendicitis (Infections and infestations) | 0 (0) | 1 (1)
Bacterial pneumonia (Infections and infestations) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tenoten for Children (N=122) | Placebo (N=118)
Hearing loss (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Eye pain (Eye disorders) | 0 (0) | 1 (1)
Functional indigestion (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 5 (5)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 4 (4)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Food intoxication (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 2 (2)
Hyperthermia (General disorders) | 2 (2) | 0 (0)
Pseudoallergy (Immune system disorders) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 2 (2) | 0 (0)
Gingivitis (Infections and infestations) | 1 (1) | 0 (0)
Laryngitis (Infections and infestations) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 2 (2) | 5 (5)
Herpes labial (Infections and infestations) | 0 (0) | 2 (2)
Pharyngitis (Infections and infestations) | 3 (3) | 2 (2)
ARI (Infections and infestations) | 7 (7) | 4 (4)
ARVI (Infections and infestations) | 14 (14) | 6 (6)
Rhinitis (Infections and infestations) | 4 (4) | 1 (1)
Runny nose (Infections and infestations) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0)
Tonsillitis (Infections and infestations) | 1 (1) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 4 (4) | 5 (5)
Hyperactivity (Nervous system disorders) | 1 (1) | 1 (1)
Tremor (Nervous system disorders) | 1 (1) | 0 (0)
Hyperexcitability syndrome (Psychiatric disorders) | 0 (0) | 1 (1)
Enuresis (Psychiatric disorders) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 2 (2) | 0 (0)
Obsessions (Psychiatric disorders) | 1 (1) | 0 (0)
Simple vocal tics (Psychiatric disorders) | 0 (0) | 1 (1)
Bronchial asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — Exacerbation of bronchial asthma
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Nose bleed (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Runny nose (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Vasomotor rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Allergic dermatitis (Skin and subcutaneous tissue disorders) | 5 (5) | 1 (1)
Pitiriasis pink (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-01-22): https://cdn.clinicaltrials.gov/large-docs/04/NCT03159104/Prot_SAP_000.pdf